CLINICAL TRIAL: NCT04462679
Title: COMMIT HIV Acceptability and Feasibility Trial
Brief Title: COMMIT HIV Trial Nepal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Possible (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Francisco (Other); Icahn School of Medicine at Mount Sinai, Department of Health Systems Design and Global Health (Unknown); Nyaya Health Nepal (Unknown); Ministry of Health and Population, Nepal (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: COMMITHIVNyaya; 1R34MH118049-01 (NIH)
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hiv
Keywords: low- and middle-income countries; mHealth; human-centered design and engineering; digital tools; Nepal; motivational interviewing; non-physician healthcare workers; community health workers; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot arm (Experimental): Mixed methods, acceptability and feasibility pilot of the COMMIT mHealth application
  Interventions: Other: COMMIT mHealth application

INTERVENTIONS:
Other: COMMIT mHealth application — We will develop Community-based mHealth Motivational Interviewing Tool (COMMIT) using iterative design and testing with frequent, structured input from the key stakeholders: community health workers (CHWs), their supervisors and youth living with HIV (YLWH).The tool will be used by community CHWs in Achham, Nepal to: 1) obtain decision-support to deliver motivational interviewing (MI) for patients in their communities, and 2) capture consented audio recordings of client interactions for review and feedback by their supervisors, allowing CHWs to maintain MI skills beyond the initial training period.

SUMMARY:
Community Healthcare Workers (CHWs), who live in the communities they serve, have the potential to reach patients who poorly engage in their care. Motivational Interviewing (MI) is a special type of interactional approach that focuses on improving the person's motivation to engage in healthy behaviors, such as keeping their clinic appointments and regularly taking medications. In this study, we will develop a mobile health tool that will assist CHWs in two tasks while they utilize MI to assist patients' engagement in care: 1) follow prompts on the mobile device to deliver MI; and 2) record consented conversations between CHWs and patients so that MI specialists can review the audiotape and provide feedback to maintain the MI skills.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for patient population: 1) having a documented HIV diagnosis, 2) living in the community health worker catchment area at the Nepal research site and , 3) having poor adherence (missed a clinic visit by more than 2 weeks, <95% adherence from visual analogue scale and/ or failed to refill their antiretroviral medications 1 week past the expected date)
2. Inclusion criteria for community health worker or a community health worker supervisor: living/working at the Nepal research site who has received motivational interviewing training as part of the intervention, and are involved directly in program implementation process.

Exclusion Criteria:

1. Exclusion criteria for patient population: includes decision from the patient to not receive care delivered by care provider at the Nepal research site or not to participate in the study
2. Exclusion criteria for a community health worker or a community health worker supervisor: includes decision not to participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-11-25 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
CD4 count | 9 months
  Individual CD4 count, measured at baseline and endline, with 350 (cells/cubic ml) as binary low/high threshold
HIV viral load | 9 months
  Individual HIV viral load count, measured at baseline and endline, with viral load suppression or >2 log drop in viral load as binary suppressed/not threshold
Self-reported HIV treatment adherence | 9 months
  Individual ART medication adherence over past month as measured by the self-reported HIV visual analogue scale (scale of 0-100%; minimum: 0%; maximum: 100%; higher scores correspond to a stronger outcome; patients asked to self-report what proportion of prescribed medications did the patient take over the past month).

SECONDARY OUTCOMES:
Application access and completion percentage | 9 months
  Frequency of community health worker accessing mobile application during study (number of times mobile application is accessed/data are entered and completed as a proportion of patients assigned for follow-up)
Patient encounter duration | 9 months
  Total amount of time spent using mobile application during patient encounter (amount of time spent in the application and at each prompt)
Application error/crash percentage | 9 months
  Frequency of mobile application displaying error messages or crashing while in use by community health workers during patient encounters (proportion of all patient encounters where an error message/application crashes occurs)

CONTACTS AND LOCATIONS:
Locations (1):
- Bayalpata Hospital, Sanfebagar-10, Achham/Province 7, Nepal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT04462679/ICF_000.pdf